CLINICAL TRIAL: NCT03896971
Title: Treatment With Thrombopoietin Mimetic Plus Immunosuppressive Therapy in Egyptian Patients With Aplastic Anaemia
Brief Title: Combination of Thrombopoietin Mimetic and Immunosuppressive Therapy in Aplastic Anaemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Safaa AA Khaled (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Safaa AA Khaled, Associate professor, Assiut University
Organization: Assiut University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKhaled19
Record Dates: First submitted 2019-03-21; First posted 2019-04-01 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Aplastic Anemia
Keywords: thrombopoietin mimetic; Egyptian; Aplastic
MeSH Terms: conditions — Anemia, Aplastic | interventions — Cyclosporine

STUDY DESIGN:
Intervention Model Description: Two groups of patients will be included one group will be treated with thrombopoietin mimetic and immunosuppressive therapy , another matched group treated with immunosuppressive therapy alone and enrolled retrospectively
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrombopoietin mimetic plus immunosuppressive therapy (Experimental): The intervention group will be given cyclosporin A plus thrombopoietin (TPO) mimetic starting with 50 mg orally daily that would be increased or decreased according to response, for 3-months. Patients will be kept on weekly follow up visits and assessed by peripheral hemogram .
  Interventions: Drug: Combination of thrombopoietin mimetic and cyclosporin A
- Immunosuppressive therapy (No Intervention): A comparative group will be collected retrospectively and treated with cyclosporin A alone as standard.

INTERVENTIONS:
Drug: Combination of thrombopoietin mimetic and cyclosporin A — This is a controlled interventional study that will be carried out in the Clinical Hematology Unit, at the Department of Internal Medicine , Assiut University Hospital. Patients will be recruited among those who attending the outpatient clinic or admitted in the unit.
  Other Names: Combination of Eltrombopag plus cyclosporin A
  Arms: Thrombopoietin mimetic plus immunosuppressive therapy

SUMMARY:
To the investigator's Knowledge this is the first study that will assess Treatment with thrombopoietin Mimetic plus immunosuppressiveTherapy in Egyptian Patients with Aplastic Anaemia.

Aim of the work :

1. To evaluate the efficacy, tolerability and toxicity of the combination of thrombopoietin mimetic and immunosuppressive therapy in Egyptian patients with AA.
2. To study the influence of this combination on patients' quality of life.
3. To access evolution to paroxysmal nocturnal hemoglobinuria (PNH), myelodysplastic syndrome , acute leukemia or development of fibrosis

DETAILED DESCRIPTION:
Aplastic anemia (AA) is a bone marrow failure syndrome that, although benign in nature, it influences patients' quality of life and carries poor prognosis.The pathophysiological basis of development of acquired AA include immune-mediated attack, inherent hematopoietic stem cell insufficiency and telomere defects. Bone marrow transplantation (BMT) is the only curative treatment for AA. Unfortunately it is unavailable for many patients due to lack of matched donors furthermore others are ineligible for BMT due to old age or co-morbid conditions. Immunosuppressive therapy was the mainstay of treatment for AA for many years, however many patients developed resistance or refractoriness. Immunosuppressive therapy was in the form of antithymocyte globulin (ATG) which gave hematologic response in nearly 50% of patients , adding cyclosporin A increases this response to 70%. Why some patients became resistant to immunosuppressive therapy ? The answer is not known.

Thrombopoietin mimetic (Eltrombopag) was firstly FDA approved for treatment of immune thrombocytopenic purpura. Numerous clinical trials proved the efficacy of anthropometric mimetic in patients with refractory severe AA, leading to its FDA approval for this group of patients. Some researchers proven the efficacy of thrombopoietin mimetic in patients with moderate aplastic anemia.

This study aimed to asses the combination of thrombopoietin mimetic and immunosuppressive therapy in patients with AA.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for treatment with thrombopoietin mimetic.
* Willing to participate in the study and signed informed consent.
* Unavailability of BMT -

Exclusion Criteria:

* Patient with inherited aplastic anemia
* Underlying immune deficiency
* Contra indication to cyclosporin A
* Endstage hepatic or renal disease
* Pregnancy and lactation

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with hematologjc response | 2-3months
  1. Platelet number ( time frame(2-3 months) : Increase plt count 20, 000 or more from baseline or independence of platelet transfusion for 2 months
  2. Hemoglobin percent (time frame (2-3 months): increase Hb by 1.5 g/dl from baseline or reduction 4 units of packed red blood cell transfusions for 2- months C) Absolute neutrophilic count response (time frame (2-3 months): increase absolute neutrophil count by 500 per microliter from baseline.
  d) Bone marrow cellularity (time frame (2-3 months): increase bone marrow cellularity from baseline

SECONDARY OUTCOMES:
Number of patients with one of the following | 2-3months
  1. Toxicity: development of toxicity leading to cessation of treatment
  2. Evolution: evolution to paroxysmal nocturnal hemoglobinuria , myelodysplastic syndrome or acute leukemia
  3. Bleeding and cytopenias that met the criteria for severe aplastic anemia and require transfusions

CONTACTS AND LOCATIONS:
Overall Officials: Safinaz Hussien, MD, Study Director — Assiut University; Sawsan A Abdelaal, M.B.B.Ch, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospital Internal Medicine Department Hematology and BMT Unit, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scheinberg P, Cooper JN, Sloand EM, Wu CO, Calado RT, Young NS. Association of telomere length of peripheral blood leukocytes with hematopoietic relapse, malignant transformation, and survival in severe aplastic anemia. JAMA. 2010 Sep 22;304(12):1358-64. doi: 10.1001/jama.2010.1376. PMID 20858879
- [Background] Frickhofen N, Kaltwasser JP, Schrezenmeier H, Raghavachar A, Vogt HG, Herrmann F, Freund M, Meusers P, Salama A, Heimpel H. Treatment of aplastic anemia with antilymphocyte globulin and methylprednisolone with or without cyclosporine. The German Aplastic Anemia Study Group. N Engl J Med. 1991 May 9;324(19):1297-304. doi: 10.1056/NEJM199105093241901. PMID 2017225
- [Background] Frickhofen N, Heimpel H, Kaltwasser JP, Schrezenmeier H; German Aplastic Anemia Study Group. Antithymocyte globulin with or without cyclosporin A: 11-year follow-up of a randomized trial comparing treatments of aplastic anemia. Blood. 2003 Feb 15;101(4):1236-42. doi: 10.1182/blood-2002-04-1134. Epub 2002 Oct 10. PMID 12393680
- [Background] Rosenfeld S, Follmann D, Nunez O, Young NS. Antithymocyte globulin and cyclosporine for severe aplastic anemia: association between hematologic response and long-term outcome. JAMA. 2003 Mar 5;289(9):1130-5. doi: 10.1001/jama.289.9.1130. PMID 12622583
- [Background] Kuter DJ. Thrombopoietin and thrombopoietin mimetics in the treatment of thrombocytopenia. Annu Rev Med. 2009;60:193-206. doi: 10.1146/annurev.med.60.042307.181154. PMID 19642221
- [Background] Desmond R, Townsley DM, Dumitriu B, Olnes MJ, Scheinberg P, Bevans M, Parikh AR, Broder K, Calvo KR, Wu CO, Young NS, Dunbar CE. Eltrombopag restores trilineage hematopoiesis in refractory severe aplastic anemia that can be sustained on discontinuation of drug. Blood. 2014 Mar 20;123(12):1818-25. doi: 10.1182/blood-2013-10-534743. Epub 2013 Dec 17. PMID 24345753